CLINICAL TRIAL: NCT06394908
Title: Registry of Minimally Invasive Urology Society for Urolithiasis Patients
Brief Title: Registry of MIUS for Urolithiasis (ReMIUS-U)
Acronym: ReMIUS-U
Status: Enrolling by invitation | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: Samsun Education and Research Hospital (Other); Gazi University (Other); Koç University (Other); Baskent University (Other); Cukurova University (Other); Ondokuz Mayıs University (Other); Muğla Sıtkı Koçman University (Other); Necmettin Erbakan University (Other); Alanya Alaaddin Keykubat University (Other); Dokuz Eylul University (Other); Hitit University (Other)
Responsible Party: Principal Investigator, Yiloren Tanidir, Associate professor, Marmara University
Other Study IDs: MIUS.2022.001
Record Dates: First submitted 2024-04-18; First posted 2024-05-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Urolithiasis; Stone, Kidney; Stone Ureter; Complication of Surgical Procedure
Keywords: Prospective studies; Registries; Urolithiasis
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Ureterolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this registry is to collect data on patients who have undergone minimally invasive treatments for urinary system stone disease, including percutaneous nephrolithotomy (PCNL), shock wave lithotripsy (SWL), semi-rigid ureterorenoscopy (URS), and flexible ureterorenoscopy (F-URS).

DETAILED DESCRIPTION:
In this project, the Minimally Invasive Urology Association urolithiasis study group aimed to collect the data of adult and pediatric urinary system stone patients treated with PCNL, SWL, URS, and F-URS in a non-randomized, observational, and prospective manner. The registry was to be conducted multi-center in Turkey.

In this project, Excel files were created and shared via Google Drive with the responsible physicians at the centers to be included in the study. Each parameter was prepared in an explanatory manner and can be readily filled out by physicians familiar with these methods. The ability to examine and modify existing data will be restricted to the worker and the database administrator. Patients' identities will not be revealed in the registry.

The collected data are summarized in three sections under the major headings below;

1. Demographics and preoperative information; Patient, disease, and treatment method demographic data, such as age, gender, height, weight, previous diseases, medications used, location, size, and hardness of urinary tract stones, the side of the stone, and the methods used for diagnosis, will be prospectively recorded for patients whose consent was obtained.
2. Data during the operation; The duration of the operation as well as the devices and methods utilized will be recorded.
3. In the postoperative period, post-treatment findings, such as stone-free status and post-treatment complications, will be documented.

A separate application to the ethics committee will be submitted for each study on the subject that will be created in the future from the multi-center, prospectively recorded data pool and on the subject that will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* To have a medical indication for urolithiasis
* Complete data of treatment and follow-up course
* Patients with consent
* Patients > 18 years-old
* Patients < 18 years-old

Exclusion Criteria:

* Missing data
* Patients without consent
* Not to have a medical indication for urolithiasis treatment
* To have a contraindication for urolithiasis treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive urolithiasis treatment without contraindication
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Operative durations of each treatment technique (PCNL, SWL, URS, F-URS) | Operation/procedure day
  The duration of the operation time
Operative radiation dosage of each treatment technique (PCNL, SWL, URS, F-URS) | Operation/procedure day
  X-ray dosage
Operative results of each treatment technique (PCNL, SWL, URS, F-URS) | Operation/procedure day
  The duration of the laser time
Postoperative results | immediately after procedure
  Postoperative estimated glomerular filtration rate (CKD Epidemiology Collaboration (CKD-EPI) equation) (mL/min/1.73 m2)
Rate of postoperative complication | up to 3 months, postoperatively
  Abnormal clinical and laboratory findings that may be seen after surgery and require additional intervention, treatment, or follow-up
Follow-up | up to 10 years
  Follow-up results of patients for recurrence of disease of residual stones, if any reoperation records.

CONTACTS AND LOCATIONS:
Overall Officials: yiloren tanidir, Assoc.Prof, Study Chair — Marmara University
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)